CLINICAL TRIAL: NCT01513408
Title: Prospective Study of the Relevance of T Lymphocytes Tumor Infiltrates CD8 and Foxp3 as a New imMUne Prognostic Biomarker in Breast Cancer Treated by NEOadjuvant Chemotherapy
Brief Title: Relevance of T Lymphocytes Tumor Infiltrates CD8 and Foxp3 as Immune Prognostic Biomarker in Breast Cancer Treated by Neo Adjuvant Chemotherapy
Acronym: PRIMUNEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2011-1SLa-01
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; CD8+; Foxp3; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD8/Foxp3 (Experimental): patient suffering from non-metastatic breast cancer
  Interventions: Other: immunohistochemical detection of lymphocytes T CD8+/Foxp3 ratio

INTERVENTIONS:
Other: immunohistochemical detection of lymphocytes T CD8+/Foxp3 ratio — For each patients included the study, a tumour block from the initial biopsy, as well as a representative block of residual tumour (area of complete tumoral regression, area of partial tumoral regression or area of unmodified residual tumour) will be chosen by the initial pathologist in each investigating centre. Once the pathologist has verified the concordance between the images observed on the blocks sent from the investigating centres, and the associated pathology reports, immunohistochemical analysis will be performed on the slides prepared from each block.

SUMMARY:
Neoadjuvant chemotherapy is standard therapy for the management of localised breast cancer, and makes it possible to evaluate tumour response. Achieving pathological complete response (pCR) after chemotherapy is the most important prognostic factor for these patients. However, patients with pCR can suffer relapse. In parallel, long-term prognosis of patients who do not achieve pCR is poorly documented, and no specific prognostic factors have been clearly identified.Preclinical and clinical studies argue for an immunogenic role of some chemotherapy regimens, such as anthracyclines, taxanes or trastuzumab. By facilitating recruitment of CD8 T-lymphocytes in the tumour bed, these agents could favourably influence antitumour immune response, partially contributing to efficacy. Conversely, tumours can promote accumulation of regulatory T-lymphocytes expressing Foxp3, thus evading anti-tumour immune response, and increased numbers of regulatory T-cells are associated with less favourable prognosis in breast cancer patients. We have previously shown that a high number of CD8 T-cells associated with low Foxp3 infiltration, as quantified by immunohistochemistry on surgical specimens, is associated with better response and better survival in breast cancer patients, independently of whether pCR was achieved, the type of chemotherapy used, and the type of breast cancer. Therefore, we propose to validate in a prospective study this immunological prognostic marker in a large cohort of patients treated with neoadjuvant chemotherapy.

ELIGIBILITY:
inclusion criteria

1. Signed informed consent
2. Social security coverage
3. Age between 18 and 80 years
4. Histologically proven breast cancer, regardless of histological type or molecular subtype (triple negative, hormone-receptor positive, HER2+++), including inflammatory forms
5. Localised breast cancer with or without axillary or subclavicular lymph node involvement
6. Absence of bone or visceral metastasis on further evaluation (bone scintigraphy, chest X-ray, abdominal echocardiography or CT scan of the thorax, abdomen and pelvic area)
7. Treatment by neoadjuvant chemotherapy (treatment protocol at physician's discretion)
8. Patient amenable to receiving adjuvant therapy (chemotherapy, radiotherapy, hormone therapy, targeted therapy)
9. Breast surgery (breast-sparing or not) planned after neoadjuvant chemotherapy

exclusion criteria

1. Metastatic breast cancer
2. Neoadjuvant radiotherapy
3. Patient not amenable to surgery
4. Ongoing therapy for any other type of cancer
5. Legal incapacity (incarceration or persons under legal guardianship)
6. Patient unable to sign the informed consent or unable to attend medical follow-up for geographical, social or mental reasons.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of inclusion up to the end of follow-up period : december 2014 (anticipated)
  Overall survival is defined as the time from inclusion date to death from any cause, or to date of last follow-up, if death does not occur.

SECONDARY OUTCOMES:
Recurrence-free survival | From inclusion up to the end of follow up period: december 2014
  Recurrence-free survival is defined as the time interval from the date of surgery to the date of first recurrence (loco-regional or metastatic) or to death (all causes). Patients alive without recurrence will be censored on the date of last follow-up.
Pathological complete response | After surgery
  Pathological complete response on the surgically resected specimen is defined as the absence of any evidence of invasive carcinoma in the breast or dissected axillary lymph nodes.
PathIm score (pathological-immunological) | From inclusion up to the end of surgery for all patients: december 2014 (anticipated)
  PathIm score (pathological-immunological)from 0 to 2, defining three patient groups with different prognoses (0 = good prognosis; 1 = intermediate prognosis; 2 = unfavourable prognosis), and defined as the sum of the pathology information regarding the extent of residual tumour according to the pAJCC score(pAJCC stage≤IIA = 0; pAJCC stage>IIA = 1), and the immunological information from the CD8/Foxp3 ratio (high CD8 AND low Foxp3 infiltration = 0, all other situations = 1)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain LADOIRE, MD, Principal Investigator — Centre Georges Francois Leclerc
Locations (1):
- CGFL, Dijon, France